CLINICAL TRIAL: NCT01980264
Title: Harmonics-based in Vivo Optical Virtual Biopsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 200903064D
Record Dates: First submitted 2013-11-03; First posted 2013-11-08 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-06

CONDITIONS: Healthy Participants With Different Skin Types and Different Ages; Diseased Participants With Different Skin Types and Different Ages; Participants Suffered From Diabetes With Different Skin Types and Different Ages
Keywords: Healthy human skin; Skin cancer; Melanoma; Basal Cell Carcinoma; Squamous Cell Carcinoma; Diabetes mellitus
MeSH Terms: conditions — Skin Neoplasms; Melanoma; Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Diabetes Mellitus | interventions — Second Harmonic Generation Microscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic imaging (Experimental): Harmonic Generation Microscopy
  Interventions: Device: Harmonic Generation Microscopy

INTERVENTIONS:
Device: Harmonic Generation Microscopy — Harmonic Generation Microscopy is a nonlinear optical microscopy.
  Other Names: HGM

SUMMARY:
The research aims to study the molecules and structures in human skin by the image formation of harmonic-based in vivo optical virtual biopsy.

DETAILED DESCRIPTION:
In the research, the investigators use the Cr:forsterite laser as the light source, and utilize the nonlinear optical microscopic system to observe human skin via in vivo detection. In this study, images of human skin tissue will be acquired by virtual section to truly evaluate the feasibility of this system in clinical application.

This research intends to conduct the following research:

1. To study the feasibility of this technology to observe melanin in the skin: As melanin is THG-bright, the technology will help to explore the distribution and change of melanin in the skin.
2. To study the capability of this technology in the early diagnosis of skin cancers, including melanoma, basal cell carcinoma, and squamous cell carcinoma: By obtaining skin images of healthy and diseased patients, we can establish an image database of normal and cancerous skin in different atages, and evaluate the efficacy of this technology for early diagnosis of skin malignancy in the future.
3. To study the ability of this technology to observe and analyze the degree of skin aging: Optical sectioning of human skin in a non-invasive in vivo manner can be used to detect the microscopic changes of skin aging and solar damage, and to find out the indicators of skin aging, so as to be used in the future to assist the therapeutic analysis of anti-skin aging treatment.
4. To study the ability of this technology to observe peripheral vasculopathy and molecular changes of microvascular structures in diabetic patients: Perform microscopic imaging on healthy and diabetes patients' skin to observe effects of structures and molecules in their skin, such as peripheral vasculopathy in diabetic patients, and the status of disease parameters, with a view to find the cause of peripheral vascular lesions and other biological information.

ELIGIBILITY:
Inclusion Criteria:

1. healthy volunteers of different skin colors and different ages
2. patients with suspected melanoma
3. patients with suspected basal cell carcinoma or squamous cell carcinoma
4. patients with diabetes mellitus

Exclusion Criteria:

1. volunteers have infectious disease
2. volunteers' skin have been infected with ulceration

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2009-08-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To noninvasively provide real-time imaging of cutaneous histopathology and molecular changes. | one year
  To observe some analyzed molecule (melanin density, HbA1c density, collagen density, etc) & structure (cell size, cell height, height of rete ridges, layer thickness, etc) parameters for different skin types & age groups. (the information above can be observed in the nonlinear images) (Cell or molecule density is defined as the cell or molecule numbers in the specific image area) (Structure can be observed and reconstructed via multiple z-depth images)

SECONDARY OUTCOMES:
To provide a diagnostic tool for diseases. | one year
  To diagnose if the analyzed pathological-related parameters (the parameters can be observed in the nonlinear images) (the pathological-related information includes cell shape, cell size, and molecular distribution (ex: chromatin, HbA1c, etc) in each single cell, etc) from Harmonic-based in Vivo Optical Virtual Biopsy can distinguish melanoma, basal cell carcinoma, squamous cell carcinoma, high & low HbA1c groups from control.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hua Liao, Doctoral, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Dermatology, National Taiwan University Hospital and College of Medicine, National Taiwan University, Taipei, Taiwan

REFERENCES:
- See also: UFO-Lab — http://ufo.ee.ntu.edu.tw/